CLINICAL TRIAL: NCT02823132
Title: Study of the Level of Mannose Binding Lectin (MBL) as a Predictor of the Onset of a Invasive Fungal Infection (IFI) During Chemo-induced Aplasia in Patients With Acute Leukemia (AL)
Brief Title: Study of the Level of a Protein Which Could Predict the Development of a Fungal Infection in Patients With Acute Leukemia
Acronym: MBL INFFONG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Goyer APJ 2013
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Acute Leukemia; Invasive Fungal Infection
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients who develop a fungal infection
  Interventions: Biological: blood sample
- patients without fungal infection
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample

SUMMARY:
The aim of this study is to investigate levels of a protein, mannose binding lectin, in patients with acute leukemia who develop or not an invasive fungal infection.

ELIGIBILITY:
Inclusion Criteria :

* persons who have provided written consent
* Patients with national health insurance cover
* Patients with malignant hemopathy who have been treated with chemotherapy able to induce profound neutropenia (PN < 500 / mm3) lasting more than 10 days.
* Patients with malignant hemopathy who have received an autologous bone marrow graft
* Patients with severe idiopathic medullar aplasia (PN < 500 / mm3) who need to be hospitalized for at least 10 consecutive days (with or without treatment with immunosuppressants)

Exclusion Criteria:

* Patients who have received an bone marrow PSC allograft (as such patients have a risk of aspergillosis, which appears in most cases after medullar recovery; they will not be included in the study).
* Patients who have received an autologous PSC graf (as the duration of neutropenia is in most cases less than 10 days).
* Patients whose neutropenia, retrospectively assessed, lasted less than 10 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with acute leukemia
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
serum level of Mannose Binding Lectin (MBL) in patients with acute leukemia | 1st day of the period of aplasia

SECONDARY OUTCOMES:
Serum levels of MBL during an episode of aplasia for both groups of patients studied | Every day except Saturday and Sunday for roughly 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France